CLINICAL TRIAL: NCT07018778
Title: Quantification of Myocardial Blood Flow in Cardiovascular Magnetic Resonance for Prediction of Fractional Flow Reserve in Coronary Catheterisation
Brief Title: CMR-derived Quantitative Perfusion for Prediction of FFR
Status: Not yet recruiting | Type: Observational
Sponsor: Kerckhoff Klinik (Other)
Responsible Party: Sponsor
Other Study IDs: AZ 107/24
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Chronic Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CCS patients: Clinical patients referred for ischaemia testing (CMR/coronary angiogram) will undergo the respective counterpart as well so that patients will have undergone both CMR and invasive testing.

SUMMARY:
Patients will undergo quantitative perfusion assessment in cardiovascular magnetic resonance imaging (dual bolus or dual sequence approach) as well as invasive coronary angiography for assessment of fractional flow reserve (FFR) including assessment of coronary flow reserve (CFR) and microcirculatory resistance (IMR).

ELIGIBILITY:
Inclusion Criteria:

* clinical indication for vasodilatator CMR or invasive coronar angiography
* capability to give informed consent

Exclusion Criteria:

* general: non-compliance, <18 years of age, pregnancy
* contraindications for CMR (non-CMR compatible device, chronic kidney disease (eGFR <30ml/min), allergies (medications)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to the clinical service for ischaemia evaluation
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Quantitative Perfusion | assessment of CMR and invasive data within 24hours
  Correlation of myocardial blood flow and perfusion reserve in CMR with invasively dervived fractional flow reserve (FFR), coronary flow reserve (CFR) and microcirculatory resistance (IMR)
Dual bolus vs dual sequence | assessment of CMR and invasive data within 24hours
  Compare both CMR-derived quantitative perfusion for prediction of FFR/CFR/IMR

SECONDARY OUTCOMES:
Strain | baseline CMR data
  Correlation of segmental perfusion and myocardial strain
Tissue characterisation | baseline CMR data
  Correlation of segmental perfusion and T1/T2/ECV/LGE
Cardiovascular Hospitalisation (CVH) | 12 months
  CVH within 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Kerckhoff Klinik, Bad Nauheim, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided